CLINICAL TRIAL: NCT00959868
Title: A Phase I Clinical Trial Assessing Intravesical Antisense Oligonucleotide Targeting Heat Shock Protein 27 for the Treatment of Superficial Bladder Cancer
Brief Title: A Study for Treatment of Superficial Bladder Cancer Using OGX-427
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vancouver Coastal Health (Other Government)
Collaborators: NCIC Clinical Trials Group (Network); Vancouver General Hospital Foundation (Unknown)
Responsible Party: Alan I. So, MD, FRCSC, Vancouver Coastal Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BL-01
Record Dates: First submitted 2009-08-13; First posted 2009-08-17 (Estimated); Last update posted 2012-02-13 (Estimated); Status verified 2012-02

CONDITIONS: Bladder Cancer
Keywords: Bladder cancer; Superficial bladder cancer (Ta or T1); Muscle invasive bladder cancer (T2); Transurethral resection; Radical cystectomy; OGX-427; Antisense oligonucleotide; Heat shock protein 27; superficial bladder tumour (Ta or T1) or CIS prior to a transurethral resection; Muscle invasive (T2) bladder cancer prior to radical cystectomy
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms; Neuronopathy, Distal Hereditary Motor, Type IIB | interventions — apatorsen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: OGX-427 — OGX-427 drug product is in 25mg/mL injection in a mannitol-phosphate buffer solution packaged to deliver at least 8mL volume from a 10mL Type I, clear glass vial (ammonium sulfate treated) with Teflon coated bromobutyl rubber stopper and sealed with an aluminum, red, flip-off over seal. The drug product is aseptically compounded and sterilized via sterile filtration prior to aseptic filling.

SUMMARY:
This is a single centre, open label, phase I dose escalation trial using a modified accelerated titration design. Patients with superficial bladder tumour (Ta or T1) or CIS and candidates for transurethral resection or muscle invasive disease (>T2) and candidates for radical cystectomy will be enrolled.

OGX-427 will be given neoadjuvantly over 8 days, followed by a transurethral resection (for superficial disease) or radical cystectomy (for muscle invasive disease).

Baseline Hsp27 levels will be determined from pre-treatment cytological samples from bladder washings and tumour biopsies performed prior to therapy.

Post-treatment PK and PD data will be determined from TUR (for Ta, T1 tumours) or radical cystectomy (for T2 tumours) specimens. A recommended phase II dose will be determined from the toxicity, tissue pK, and percentage of Hsp27 knockdown. Effects of treatment on Hsp27 client protein levels and apoptotic index will also be evaluated.

Evaluation during protocol treatment will take place to assess toxicity. Assessments will occur on various visits as per Evaluation Schedule. Adverse event evaluation based on NCI CTCAEv3.0. For quality of life assessment during treatment, the EORTC QLC-BLS24 will be used before first treatment (day 1) and prior to surgery (TURBT or radical cystectomy). The Day 1 QOL assessment will serve as baseline.

After removal from protocol treatment, all subjects will be followed for toxicity related to study drug for 30 days.

After the study, subjects will be followed according to standard of care. Follow-up for tumour recurrence or superficial tumours will be assessed every three months by cystoscopic examination for two years, then every six months for the next two years, and then yearly thereafter.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age must be > 18
2. Histologic evidence of bladder cancer (superficial or muscle invasive) or

   CIS as evidenced by:
   * Patients presenting with superficial tumours and unknown pathological stage will have in-clinic bladder washings (performed cystoscopically) and biopsy (cup biopsy).
   * Patients with recurrent superficial disease (Ta or T1) and tissue that is available for baseline studies (i.e. tissue from previous transurethral resection stored in paraffin blocks) will be eligible for trial without requiring cytology or biopsy.

     * Patients with previously diagnosed T1 tumours and requiring re-resection of bladder tumour will be eligible if tissue from the original TURBT is available for baseline studies.
     * Patients presenting as muscle invasive (>T2) disease will be eligible if they are candidates for radical cystectomy and if baseline tissue from initial resections is available for baseline studies
3. No intravesical therapies within the previous 6 months
4. No evidence of metastatic disease as determined by physical exam, CT scan or chest- x-ray, where indicated.
5. ECOG status must be 0, 1, or 2
6. Laboratory requirements (within 7 days of treatment):

   * negative urine cultures
   * Absolute neutrophils count> 1.5 x 109 cells/L, and platelets count> 100 x 109/L,
   * Total bilirubin < 1.5 x upper normal limit (ULN), AST and/or ALT < 1.5 x ULN, alkaline phosphatase < 1.5 x ULN, and serum creatinine < 1.5 x ULN.
   * PTT and INR, within normal limits
7. Patient must be able to complete the quality of life questionnaires in either English or French
8. Patients must provide written informed consent.

Exclusion Criteria:

1. Patients with "indeterminate" or "negative" results from biopsy or cytology will be ineligible for the trial.
2. Patients taking warfarin or Coumadin anticoagulation therapy or who have a bleeding disorder. NOTE: Patients who require anticoagulation therapy while on study will be removed from study treatment.
3. Pregnant or lactating women
4. Patients not accessible for follow-up
5. Patients with an active urinary tract infection, upper tract urothelial tumors, active infection including tuberculosis, concurrent febrile illness or impaired immune response from any cause
6. Patients with contraindication to spinal or general anesthesia required for a transurethral resection or radical cystectomy
7. Recent (<14 days) urethral trauma or inability to perform catheterization or cystoscopy safely
8. Patients known to have a serious illness or medical condition that would impair protocol treatment delivery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
To define the maximum tolerated dose (MTD) of OGX-427 administered as an intravesical instillation. | One year
  The study medication will be escalated according to a fixed dose escalation plan. Three subjects will be treated per cohort. If one of the three subjects experiences a DLT, three additional subjects will be treated at that dose level (i.e. maximum of 6 subjects per cohort)
To define the dose-limiting toxicities (DLTs) of OGX-427 administered as an intravesical instillation. | one year
  The study medication will be escalated according to a fixed dose escalation plan. Three subjects will be treated per cohort. If one of the three subjects experiences a DLT, three additional subjects will be treated at that dose level(i.e. maximum of 6 subjects per cohort)

SECONDARY OUTCOMES:
To determine the toxicity profile of OGX-427 when administered intravesically. | One year
To measure evidence of OGX-427 effect on expression of Hsp27. | one year
To determine the bladder PK and PD profile of OGX-427 after intravesical administration. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Alan I So, MD, FRCSC, Principal Investigator — Vancouver Coastal Health
Locations (1):
- The Prostate Centre at Vancouver General Hospital, Vancouver, British Columbia, Canada